CLINICAL TRIAL: NCT04106791
Title: Evaluation of Closed-loop Control of Vasopressor Infusion in Critically Ill Patients: A Pilot Study
Brief Title: Computer Assisted Vasopressor Titration in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P2018276
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Closed-Loop Communication
MeSH Terms: conditions — Teach-Back Communication

STUDY DESIGN:
Intervention Model Description: SINGLE GROUP ASSIGNMENT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop (Experimental): Pilot study: one single group of 10 ICU patients.
  Interventions: Device: closed-loop system for vasopressor administration

INTERVENTIONS:
Device: closed-loop system for vasopressor administration — The closed-loop system' goal is to keep MAP within 5 mmHg of the predefined target MAP.

SUMMARY:
The purpose of this pilot study is to evaluate the performance of a novel closed-loop (automated) vasopressor administration system that delivers norepinephrine using feedback from standard operating room hemodynamic monitor (EV1000 Monitor-Flotrac Edwards Lifesciences, IRVINE, USA) in 10 to 12 critically ill patients in the intensive care unit.

DETAILED DESCRIPTION:
The investigators have developed an automated closed-loop system for vasopressor administration . They will test it in critically ill patients. The investigators want to demonstrate that the closed-loop system can maintain mean arterial pressure ( MAP) within a very narrow range (within +/- 5 mmHg of the predefined MAP target) for more than 85 % of the treatment time.

The Investigators have shown this to be the case in simulation studies and in-vivo animal studies and in surgical patients but not yet in the Intensive care unit (ICU). Investigators will recruit 10 to 12 ICU patients equipped with a mini-invasive cardiac output monitoring and under continuous norepinephrine infusion.

These patients will typically include: septic patients, neuro ICU patients, ARDS patients, trauma patients or postoperative patients.

The target MAP will be determined by the ICU physician in charge of the patient.

Fluids will be given standard of care. The closed loop (automated) system will use an infusion pump (Q-Core and chemyx pump) and a controller (a computer run index and algorithm developed by Sironis) to make frequent, regular and accurate adjustments of vasopressor (norepinephrine)

The goal is to register a period of two hours of closed-loop control of MAP.

ELIGIBILITY:
Inclusion Criteria:

- ICU patients under norepinephrine administration and equipped with a advanced hemodynamic monitoring device

Exclusion Criteria:

* Subjects under 18 years of age
* Subjects not requiring cardiac output monitoring or an arterial line
* Subject with Atrial Fibrillation
* Subjects who are pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of case Time in target (MAP within 5 mmHg of the predetermined MAP target). | 48 hours post-admission in the intensive care
  The primary outcome will be the percentage of case time in target

SECONDARY OUTCOMES:
Percentage of case Time in hypotension (MAP <5 mmHg of the chosen target) | 48 hours post-admission in the intensive care
  Percentage of case Time in hypotension (MAP <5 mmHg of the chosen target)
Percentage of case time with MAP >5 mmHg of the chosen target with vasopressor still running. | 48 hours post-admission in the intensive care
  Percentage of case time with MAP >5 mmHg of the chosen target with vasopressor still running.
Amount of vasopressors received | 48 hours post-admission in the intensive care
  Amount of vasopressors received
Number of vasopressor modifications over the treatment time | 48 hours post-admission in the intensive care
  Number of vasopressor modifications (increase or decrease infusion rate) over the treatment time
Limitations of the closed-loop system | 48 hours post-admission in the intensive care
  Number of errors, malfunction of the system during the treatment time

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre J MD, PhD, Principal Investigator — ERASME
Locations (1):
- Erasme, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No